CLINICAL TRIAL: NCT06536907
Title: The Effect of Decompression on Histologic Diagnoses of Cystic Jaw Lesions
Brief Title: Decompression of Odontogenic Cysts
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Altay, Associate Professor, Akdeniz University
Other Study IDs: 70904504/553
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Odontogenic Cysts; Keratocysts of the Jaw; Cysts Dental; Pathology
Keywords: biopsy; diagnosis; keratocysts; odontogenic cysts; oral pathology; surgical decompression
MeSH Terms: conditions — Odontogenic Cysts; Radicular Cyst; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this case-control study is to evaluate the effects of decompression of cystic jaw lesions by means of comparing pre- and post-decompression histologic findings.

The main question it aims to answer is:

Does decompression of cystic jaw lesions alter the histologic diagnosis?

A retrospective analysis was performed based on the comparison of initial and final histologic diagnoses of patients with an odontogenic cystic lesion, that was surgically treated with decompression followed by a definitive surgery.

DETAILED DESCRIPTION:
The study included patients with a histologic diagnosis of an odontogenic cystic lesion, that was surgically treated with decompression followed by a definitive surgery. The study was carried out retrospectively by means of evaluating records, surgical and histologic reports of patients. Pre- and post-decompression histologic findings were compared in effort to understand if decompression leads to alteration in histologic character and change in diagnoses of lesions.

ELIGIBILITY:
Inclusion Criteria:

* To have an initial diagnosis of an odontogenic cystic jaw lesion confirmed with an incisional biopsy.
* The patients must have undergone decompression and, enucleation or enucleation and peripheral ostectomy after decompression period.

Exclusion Criteria:

* Previously treated patients
* The patients with missing information in medical and/or dental records
* The patients who did not adhere to follow-up protocol

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included patients with a histologic diagnosis of an odontogenic cystic lesion, that was surgically treated with decompression followed by a definitive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in histologic diagnosis following decompression (yes/no) | A decompression period ranging between 2 and 15 months
  A comparison will be made between the initial histologic diagnosis and post-decompression definitive histologic diagnosis of the cystic jaw lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rajendra Santosh AB. Odontogenic Cysts. Dent Clin North Am. 2020 Jan;64(1):105-119. doi: 10.1016/j.cden.2019.08.002. Epub 2019 Oct 18. PMID 31735221
- [Result] Wakolbinger R, Beck-Mannagetta J. Long-term results after treatment of extensive odontogenic cysts of the jaws: a review. Clin Oral Investig. 2016 Jan;20(1):15-22. doi: 10.1007/s00784-015-1552-y. Epub 2015 Aug 8. PMID 26250795
- [Result] Oliveros-Lopez L, Fernandez-Olavarria A, Torres-Lagares D, Serrera-Figallo MA, Castillo-Oyague R, Segura-Egea JJ, Gutierrez-Perez JL. Reduction rate by decompression as a treatment of odontogenic cysts. Med Oral Patol Oral Cir Bucal. 2017 Sep 1;22(5):e643-e650. doi: 10.4317/medoral.21916. PMID 28809378
- [Result] Mohanty S, Dabas J, Verma A, Gupta S, Urs AB, Hemavathy S. Surgical management of the odontogenic keratocyst: A 20-year experience. Int J Oral Maxillofac Surg. 2021 Sep;50(9):1168-1176. doi: 10.1016/j.ijom.2021.02.015. Epub 2021 Mar 2. PMID 33663899
- [Result] Anavi Y, Gal G, Miron H, Calderon S, Allon DM. Decompression of odontogenic cystic lesions: clinical long-term study of 73 cases. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Aug;112(2):164-9. doi: 10.1016/j.tripleo.2010.09.069. Epub 2010 Dec 30. PMID 21194990
- [Result] Pogrel MA, Jordan RC. Marsupialization as a definitive treatment for the odontogenic keratocyst. J Oral Maxillofac Surg. 2004 Jun;62(6):651-5; discussion 655-6. doi: 10.1016/j.joms.2003.08.029. PMID 15170272
- [Result] Schlieve T, Miloro M, Kolokythas A. Does decompression of odontogenic cysts and cystlike lesions change the histologic diagnosis? J Oral Maxillofac Surg. 2014 Jun;72(6):1094-105. doi: 10.1016/j.joms.2013.12.028. Epub 2014 Jan 15. PMID 24576437
- [Result] Allon DM, Allon I, Anavi Y, Kaplan I, Chaushu G. Decompression as a treatment of odontogenic cystic lesions in children. J Oral Maxillofac Surg. 2015 Apr;73(4):649-54. doi: 10.1016/j.joms.2014.10.024. Epub 2014 Oct 31. PMID 25631867
- [Result] Berretta LM, Melo G, Mello FW, Lizio G, Rivero ERC. Effectiveness of marsupialisation and decompression on the reduction of cystic jaw lesions: a systematic review. Br J Oral Maxillofac Surg. 2021 Dec;59(10):E17-E42. doi: 10.1016/j.bjoms.2021.03.004. Epub 2021 Mar 23. PMID 34749963
- [Result] August M, Faquin WC, Troulis MJ, Kaban LB. Dedifferentiation of odontogenic keratocyst epithelium after cyst decompression. J Oral Maxillofac Surg. 2003 Jun;61(6):678-83; discussion 683-4. doi: 10.1053/joms.2003.50137. PMID 12796876
- [Result] Nakamura N, Mitsuyasu T, Mitsuyasu Y, Taketomi T, Higuchi Y, Ohishi M. Marsupialization for odontogenic keratocysts: long-term follow-up analysis of the effects and changes in growth characteristics. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Nov;94(5):543-53. doi: 10.1067/moe.2002.128022. PMID 12424446
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Bull World Health Organ. 2007 Nov;85(11):867-72. doi: 10.2471/blt.07.045120. PMID 18038077
- [Result] Castro-Nunez J. Decompression of Odontogenic Cystic Lesions: Past, Present, and Future. J Oral Maxillofac Surg. 2016 Jan;74(1):104.e1-9. doi: 10.1016/j.joms.2015.09.004. Epub 2015 Sep 21. PMID 26428611
- [Result] Mustansir-Ul-Hassnain S, Chandavarkar V, Mishra MN, Patil PM, Bhargava D, Sharma R. Histopathologic and immunohistochemical findings of odontogenic jaw cysts treated by decompression technique. J Oral Maxillofac Pathol. 2021 May-Aug;25(2):272-278. doi: 10.4103/0973-029X.325126. Epub 2021 Aug 31. PMID 34703121
- [Result] Castro-Nunez J, Wiscovitch AG, Porte JP, Wiscovitch J, Rivera B, Guerrero LM. Does active decompression of odontogenic keratocyst change the histologic diagnosis? Oral Maxillofac Surg. 2022 Jun;26(2):291-298. doi: 10.1007/s10006-021-00994-4. Epub 2021 Jul 29. PMID 34324108
- [Result] Awni S, Conn B. Decompression of keratocystic odontogenic tumors leading to increased fibrosis, but without any change in epithelial proliferation. Oral Surg Oral Med Oral Pathol Oral Radiol. 2017 Jun;123(6):634-644. doi: 10.1016/j.oooo.2016.12.007. Epub 2016 Dec 30. PMID 28377093
- [Result] Rodu B, Tate AL, Martinez MG Jr. The implications of inflammation in odontogenic keratocysts. J Oral Pathol. 1987 Nov;16(10):518-21. doi: 10.1111/j.1600-0714.1987.tb00684.x. PMID 3127567
- [Result] Zhang L, Liu SL, Ye WM, Zheng J. STAT3 is a key pathway in primary intraosseous squamous cell carcinoma arising from an odontogenic keratocyst. Am J Transl Res. 2015 Oct 15;7(10):1860-9. eCollection 2015. PMID 26692930